CLINICAL TRIAL: NCT04956406
Title: The Effect of Motivational Interviewing on Self-Management in Adult Kidney Transplant Recipients Versus Routine Care
Brief Title: Motivational Interviewing for Adult Kidney Transplant Recipients
Acronym: MIAKTR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Cigdem Erdem, Research Asistant, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0000
Record Dates: First submitted 2021-06-25; First posted 2021-07-09 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Motivational Interviewing; Adult; Kidney Transplantation; Self-Management; Treatment Adherence; Medication Adherence; Patient Outcome Assessment
Keywords: Motivational Interviewing; Recipient; Kidney Transplantation; Self-Management
MeSH Terms: conditions — Treatment Adherence and Compliance; Medication Adherence | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant
Masking Description: The statistician will be blinded to avoid evaluator bias.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIAKTR (Experimental): MIAKTR is an acronym that defines Motivational Interviewing for Adult Kidney Transplant Recipients
  Interventions: Behavioral: Motivational Interviewing for Adult Kidney Transplant Recipients
- Control Group (Active Comparator): routine care
  Interventions: Other: Routine care

INTERVENTIONS:
Behavioral: Motivational Interviewing for Adult Kidney Transplant Recipients — Motivational interviewing with individual sessions are planned to be conducted 3 times. Planned motivational interviews will be implemented the intervention group who are within 3th month, 4th month, 5th month and 6th month. Motivational interviewing will planned last 15-30 minutes with an interval of 10 days. The first interview will be performed face-to-face at the transplant outpatient clinic and the second and third ones will be phone interviews
  Arms: MIAKTR
Other: Routine care — The control group will be provided with routine care( face-to-face care standard training) by the nurse educator at the transplant outpatient clinic.
  Arms: Control Group

SUMMARY:
Purpose: This study aimed to determine the effect of motivational interviewing on self-management of treatment regimen, medication adherence, and patient outcomes in adult kidney transplant recipients between 3 months and 6 months after kidney transplant in the transplant outpatient clinic.

Design: The research is a single-centered, single-blind, parallel and 1:1 randomized active comparative experimental study.

Method: A total of 80 individuals, of the 40 in the control group and 40 in the intervention group, will be included in the study. Motivational interview sessions for the intervention group will be held 3 times between 15-30 minutes with an interval of 10 days. The control group will be given routine care (approximately 1 hour of face-to-face standard training) by the nurse educator. Within the research pattern, intervention and control groups will be applied pre-test at the first interview and post test after one month. In addition, follow-up test will be performed 3th month. The data will be obtained using the Self-Management Scale in Kidney Transplant Recipients, Visual Analog Scale (VAS) for self-care and VAS for medication adherence. In the study, Standard Protocol Items: Recommendations for Interventional Trials- SPIRIT(2013) and CONSORT 2010 (Consolidated Standards of Reporting Trials) were used.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study,
* aged ≥18 years old
* 3-6 months after kidney transplant
* Speaking, reading and writing in Turkish
* Having a mobile phone

Exclusion Criteria:

* Request to leave work

Removing Criteria:

* Development of rejection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Self-management scale | Change from Baseline Self Management at 3 months
  The scale Turkish version includes 13 items, and it is likert type with 4 steps. Scale items are scored as 1 "never applied", 2 "applied slightly", 3 "applied very often" and 4 "fully applied". It is recommended to perform calculation based on the item mean scores instead of an overall mean. The lowest possible score obtained from each item and sub-scale is 1 and the highest possible score is 4. The scale has no cutoff points and reversed items.
VAS for medication adherence | Change from Baseline VAS for Medication Adherence at 3 months
  Medication adherence will be evaluated with self reported scale the visual analog scale ranges from 0 to 100. Rating will be of 0 "taken no medications" to 100 "taken medications perfectly". A score different from 100 will be considered a non adherence
VAS for self care | Change from Baseline VAS for self care at 3 months
  The rating will be done as 0-100. 0: "I cannot provide my own care".100:"I am able to provide my own care".

SECONDARY OUTCOMES:
Glomerular Filtration Rate (GFR) | Change from Baseline GFR at 3 months
  official measurements made by the hospital
Serum Creatinine | Change from Baseline Serum Creatinine at 3 months
  official measurements made by the hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No